CLINICAL TRIAL: NCT03547804
Title: A Prospective, Single-center, One-arm Clinical Study of Apatinib Combined With Chemotherapy for Pretreated Patients With Advanced Small Cell Lung Cancer
Acronym: MK 01
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The First Hospital of Jilin University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: K2018012
Record Dates: First submitted 2018-05-24; First posted 2018-06-06 (Actual); Last update posted 2020-12-01 (Actual); Status verified 2020-09

CONDITIONS: Small-cell Lung Cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — apatinib; Drug Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- experimental arm (Experimental): apatinib 500 mg qd;The dose was later reduced from 500 mg to 250 mg per day based on a recommendation of the principal investigator to reduce the adverse events.Chemotherapeutic agents are limited to irinotecan or docetaxel alone.
  Interventions: Drug: Apatinib; Drug: chemotherapy

INTERVENTIONS:
Drug: Apatinib — 500 mg qd/250mg
Drug: chemotherapy — Chemotherapeutic agents are limited to irinotecan or docetaxel alone.

SUMMARY:
At present, with the increasing intensities of the tobacco industry and air pollution in China, the incidence and mortality of lung cancer have become the most important issue that threatens human health.Over the past two decades, the treatment of SCLC still stays in the mode of treatment based on radiotherapy and chemotherapy.

This is a prospective, single-center, one-arm clinical study designed to evaluate the efficacy and safety of apatinib plus chemotherapy for second-line and above treatment of advanced SCLC.

30 patients will receive apatinib 500mg qd orally, if the patient has a grade 3/4 adverse reaction during apatinib treatment, it can be reduced to apatinib 250mg qd orally.The dose was later reduced from 500 mg to 250 mg per day based on a recommendation of the principal investigator to reduce the adverse events. Chemotherapeutic agents are limited to irinotecan or docetaxel alone.The primary outcome endpoint was progression-free survival

ELIGIBILITY:
Inclusion Criteria:

1, male or female patients: 18-75 years old;

2. ECOG performance status score: 0~2 points;

3, pathological examination specifically for small cell lung cancer

4. Expected survival period ≥12 weeks;

5. The normal function of major organs, that is, the relevant inspection indicators within the first 14 days of randomness, meet the following requirements:

1) Blood tests:

a) Hemoglobin ≥ 90 g/L (without transfusion in 14 days); b) Neutrophil count ≥ 1.5×109/L; c) Platelet count ≥ 100×109/L; 2) Biochemical check:

1. total bilirubin ≤ 1.5 x ULN (upper limit of normal value);
2. serum alanine aminotransferase (ALT) or serum aspartate aminotransferase (AST) ≤ 2.5 × ULN; if liver metastases, ALT or AST ≤ 5 × ULN;
3. Serum creatinine < 1.5 times the upper limit of normal; Endogenous creatinine clearance ≥ 50 ml/min (Cockcroft-Gault formula); 3) Assessment of cardiac Doppler ultrasound: Left ventricular ejection fraction (LVEF) ≥ 50%.

   6. Women of childbearing age must have a pregnancy test (serum or urine) within 7 days prior to enrollment, and the result is negative, and they are willing to use appropriate methods of contraception during the trial and within 8 weeks of the last administration of the test drug. For males, consent must be given for contraception or surgical sterilization within 8 weeks of the test period and the last administration of the test drug;

   7. Subjects have completely healed after surgery and no bleeding tendency;

   8. Good compliance, family members agree to follow the survival follow-up;

   9. Sign the informed consent form.

   Exclusion Criteria:
   1. in the past or at the same time suffering from other malignant tumors,
   2. participated in other drug clinical trials within four weeks;
   3. has a variety of factors that affect oral medication (such as inability to swallow, chronic diarrhea, and intestinal obstruction);

   4. There is a history of bleeding, and any serious grading within 4 weeks prior to screening has reached 3 degrees or more in CTCAE 4.0;

   5. Pre-screening patients with symptomatic central nervous system metastasis or history of central nervous system metastasis;

   6, patients who undergo chest radiotherapy during the first-line treatment can be enrolled in the group;

   7. People with high blood pressure who cannot be well controlled by single antihypertensive drugs (systolic blood pressure > 140 mmHg, diastolic blood pressure> 90 mmHg); patients with a history of unstable angina; newly diagnosed angina in the first 3 months before screening or myocardial infarction within 6 months prior to screening; arrhythmia (including QTcF: male ≥450 ms , ≥ 470 ms for females) long-term use of antiarrhythmic drugs and New York Heart Association grade ≥ grade II cardiac insufficiency;

   8, urine prompts urinary protein ≥ ++ and confirmed 24-hour urinary protein quantification> 1.0 g;

   9, combined with anastomotic leakage, duodenal stump fistula, pancreatic fistula or anastomotic stenosis and other serious postoperative complications;

   10. Long-term unhealed wounds or incompletely-healed fractures;

   11. Imaging shows that the tumor has invaded an important blood vessel or the investigator judged that the patient's tumor had a high risk of invading vital blood vessels and causing fatal bleeding during treatment;

   12, abnormal coagulation, bleeding tendency (14 days before randomization must meet: in the absence of resistance In the case of coagulants, the INR is within the normal range; Patients treated with anticoagulants or vitamin K antagonists such as warfarin, heparin, or the like; International normalized ratio (INR) ≤ 1.5 for prothrombin time Under the premise that small doses of warfarin (1 mg orally, once daily) or low dose aspirin (with daily dose not exceeding 100 mg) are allowed for prophylactic purposes;

   13. Incidence of arteriovenous/venous thromboembolism within the first year of screening, such as cerebrovascular accident (including transient ischemic attack), deep venous thrombosis (except for venous thrombosis due to venous catheterization in previous chemotherapy) ) and pulmonary embolism;

   14. For female subjects: Surgical sterilization, postmenopausal patients, or agree to use a medically approved contraceptive measure during study treatment and within 6 months of the end of the study treatment period; prior to study enrollment Serum or urine pregnancy tests must be negative within 7 days and must be non-lactating. Male subjects: Should be surgically sterilized, or agree to use a medically-accepted contraceptive treatment during study treatment and within 6 months of the end of the study treatment period;

   15. In the past, there was abnormal thyroid function. Even in the case of drug therapy, thyroid function could not be maintained within the normal range.

   16. Those who have a history of abuse of psychotropic substances and are unable to get rid of or have mental disorders;

   17. Has a history of immunodeficiency, or has other acquired, congenital immunodeficiency disorders, or has a history of organ transplantation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2018-05-31 (Actual); Primary Completion 2019-10-25 (Actual); Study Completion 2020-09-01 (Actual)

PRIMARY OUTCOMES:
PFS | 1 year
  Progression-free survival

SECONDARY OUTCOMES:
OS | 5 years
  Overall survival
AEs | 1 year
  Adverse events
DCR | 1 year
  Disease Control Rate
ORR | 1 year
  Objective Response Rate

CONTACTS AND LOCATIONS:
Locations (1):
- The First Hospital Of Jilin University, Changchun, Jilin, China

REFERENCES:
- [Background] Li J, Qin S, Xu J, Xiong J, Wu C, Bai Y, Liu W, Tong J, Liu Y, Xu R, Wang Z, Wang Q, Ouyang X, Yang Y, Ba Y, Liang J, Lin X, Luo D, Zheng R, Wang X, Sun G, Wang L, Zheng L, Guo H, Wu J, Xu N, Yang J, Zhang H, Cheng Y, Wang N, Chen L, Fan Z, Sun P, Yu H. Randomized, Double-Blind, Placebo-Controlled Phase III Trial of Apatinib in Patients With Chemotherapy-Refractory Advanced or Metastatic Adenocarcinoma of the Stomach or Gastroesophageal Junction. J Clin Oncol. 2016 May 1;34(13):1448-54. doi: 10.1200/JCO.2015.63.5995. Epub 2016 Feb 16. PMID 26884585
- [Background] Huang L, Wei Y, Shen S, Shi Q, Bai J, Li J, Qin S, Yu H, Chen F. Therapeutic effect of apatinib on overall survival is mediated by prolonged progression-free survival in advanced gastric cancer patients. Oncotarget. 2017 Apr 25;8(17):29346-29354. doi: 10.18632/oncotarget.12897. PMID 27793017
- [Background] Kim KL, Suh W. Apatinib, an Inhibitor of Vascular Endothelial Growth Factor Receptor 2, Suppresses Pathologic Ocular Neovascularization in Mice. Invest Ophthalmol Vis Sci. 2017 Jul 1;58(9):3592-3599. doi: 10.1167/iovs.17-21416. PMID 28715845
- [Background] Li F, Zhu T, Cao B, Wang J, Liang L. Apatinib enhances antitumour activity of EGFR-TKIs in non-small cell lung cancer with EGFR-TKI resistance. Eur J Cancer. 2017 Oct;84:184-192. doi: 10.1016/j.ejca.2017.07.037. Epub 2017 Aug 17. PMID 28822888
- [Background] Wu F, Zhang S, Gao G, Zhao J, Ren S, Zhou C. Successful treatment using apatinib with or without docetaxel in heavily pretreated advanced non-squamous non-small cell lung cancer: A case report and literature review. Cancer Biol Ther. 2018 Mar 4;19(3):141-144. doi: 10.1080/15384047.2017.1414757. Epub 2018 Jan 15. PMID 29261000